CLINICAL TRIAL: NCT07007650
Title: Effects of Different Concentrations of Ropivacaine on Prolonged Labor Analgesia
Brief Title: Effects of Ropivacaine Concentrations on Prolonged Labor Analgesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Jinjiang Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Fei Jia, Director of Anesthesiology Department, Chengdu Jinjiang Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202312
Record Dates: First submitted 2025-05-26; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Labor Analgesia; Prolonged; Ropivacaine; Concentration
Keywords: Labor Analgesia; Ropivacaine Concentration; Prolonged Pain; Maternal-Neonatal Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind design is a research method aimed at eliminating bias between participants and researchers. In this design, participants are randomly assigned to different intervention groups (such as different concentrations of ropivacaine), and neither the participants nor the researchers responsible for evaluating the results are aware of the specific group allocations. This ensures the objectivity and reliability of the research findings, avoiding the influence of subjective expectations or observational biases on data interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high concentration ropivacaine group (Experimental): The combination of 0.12% ropivacaine and 0.5 μg/ml sufentanil
  Interventions: Drug: High-concentration Ropivacaine
- Low concentration ropivacaine group. (Active Comparator): The combination of 0.1% ropivacaine and 0.5 μg/ml sufentanil
  Interventions: Drug: Low concentration ropivacaine group

INTERVENTIONS:
Drug: High-concentration Ropivacaine — After the first pump fluid is depleted, switch to 0.12% ropivacaine to continue labor analgesia.
  Arms: high concentration ropivacaine group
Drug: Low concentration ropivacaine group — After the first pump fluid is depleted, switch to 0.12% ropivacaine to continue labor analgesia.
  Arms: Low concentration ropivacaine group.

SUMMARY:
With the changes in medical models and improvements in people's quality of life, parturients have higher demands for childbirth, making the alleviation and elimination of labor pain an important aspect of modern obstetrics. Intrathecal labor analgesia has been widely adopted in clinical practice to relieve pain. However, current studies mainly focus on parturients who are just beginning to receive labor analgesia, while for those experiencing prolonged analgesia, medical institutions still use traditional formulations, lacking relevant guidelines or expert consensus. In such cases, prolonged waiting and anxiety may lower the pain tolerance of parturients, leading to an increased need for higher concentrations of local anesthetics. To address this clinical gap, this study aims to explore the effects of different concentrations of ropivacaine in prolonged labor analgesia and has designed a prospective randomized controlled trial (RCT) to provide evidence for improving the analgesic regimen for this group of parturients.

DETAILED DESCRIPTION:
Background:

With changes in medical models and improvements in quality of life, parturients have higher expectations for childbirth, making the alleviation and elimination of labor pain an important aspect of modern obstetrics. Intrathecal labor analgesia is widely used in clinical practice to relieve labor pain. However, studies on prolonged labor analgesia, especially following the replacement of the first analgesic pump, are scarce. Medical institutions often continue to use traditional analgesic formulations without relevant guidelines or expert consensus. Prolonged analgesia may reduce pain tolerance in parturients, possibly necessitating adjustments in local anesthetic concentration to improve analgesic effectiveness. Given the clinical research gap, this study aims to explore the effects of different concentrations of ropivacaine on prolonged labor analgesia and its impact on maternal and neonatal safety.

Objective:

To investigate the effects and maternal-neonatal safety of using different concentrations of ropivacaine for prolonged labor analgesia, providing clinical evidence for optimizing labor analgesia regimens.

Methods:

This single-center prospective randomized controlled study will collect clinical data from parturients receiving labor analgesia at Chengdu Jinjiang District Maternal and Child Health Hospital from May to August 2025. Participants meeting the inclusion and exclusion criteria will be included. Following the replacement of the first analgesic pump, parturients will be randomly assigned to receive one of two ropivacaine concentration regimens (Group H: 0.12% ropivacaine; Group N: 0.1% ropivacaine). Data collection will include demographic information, pain scores, labor-related parameters, neonatal outcomes, and adverse reactions.

Interventions:

1. Group H: 0.12% ropivacaine + 0.5µg/ml sufentanil
2. Group N: 0.1% ropivacaine + 0.5µg/ml sufentanil Following the replacement of the first analgesic pump, parturients will receive the respective ropivacaine concentration formulation, with pain relief effects and labor-related indicators assessed at specified intervals.

Primary Outcome:

Pain scores at different time points (T0: at pump replacement; T1: 0.5 hours after pump replacement; T2: 1 hour after pump replacement; T3: at full cervical dilation or during transition to cesarean section).

Secondary Outcomes:

1. Labor-related indicators: Duration of first, second, and third stages of labor, blood loss, rate of instrumental delivery, mode of delivery (vaginal/cesarean).
2. Neonatal indicators: Neonatal weight, Apgar scores at 1 minute, 5 minutes, and 10 minutes.
3. Adverse reactions: Hypotension, nausea/vomiting, intrapartum fever (T≥38.0℃).

Hypothesis:

Different concentrations of ropivacaine for prolonged intrathecal labor analgesia will have varying effects on pain control and maternal-neonatal safety, with higher concentration ropivacaine (0.12%) likely being more effective in pain relief, while both concentrations are expected to show no significant difference in maternal and neonatal safety.

Ethics Approval:

This study has received approval from the ethics committee of Chengdu Jinjiang District Maternal and Child Health Hospital (Approval Number: 202312). All participants must sign an informed consent form to ensure the respect of participant rights and data confidentiality. The study will strictly adhere to relevant ethical standards and legal regulations to protect participant safety and privacy.

Funding:

This study is funded by the following projects:

1. Chengdu Medical Research Project (No. 2023465)
2. Chengdu Medical Research Project (No. 2022548)
3. Chengdu Medical Research Project (No. 2023304)

ELIGIBILITY:
Inclusion Criteria:

1. ASA II
2. Age ≥ 18 years
3. Singleton pregnancy
4. No contraindications for epidural puncture and voluntarily accepting labor analgesia
5. Maternal participants changing the first pump fluid

Exclusion Criteria:

1. Contraindications for epidural labor analgesia
2. Serious heart, brain, liver, or kidney diseases
3. Mental abnormalities
4. Neurological diseases
5. Maternal request for management of breakthrough pain before changing the pump fluid

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to women who are planning a vaginal delivery and voluntarily accepting labor analgesia.
Enrollment: 100 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | From pump replacement to the end of labor analgesia.
  The pain will be assessed using the Visual Analog Scale (VAS) at four time points:
  T0 (at the time of pump fluid change) T1 (0.5 hours after the pump fluid change) T2 (1 hour after the pump fluid change) T3 (when full cervical dilation is achieved/in case of emergency cesarean section).

SECONDARY OUTCOMES:
Modified Bromage score | From pump replacement to the end of labor analgesia.
  The level of motor blockade will be assessed using the Modified Bromage Score at four time points:
  T0 (at the time of pump fluid replacement) T1 (0.5 hours after the pump fluid replacement) T2 (1 hour after the pump fluid replacement) T3 (at full cervical dilation/in case of emergency cesarean section)
Mode of delivery | At the end of delivery
  The mode of delivery will be recorded (vaginal birth/cesarean section).
Neonatal Apgar score | 10 minutes after the delivery of the fetus
  The Apgar Score will be recorded for the newborn at 1 minute, 5 minutes, and 10 minutes after delivery.
nausea and vomiting questionnaire | From pump replacement to the end of labor analgesia.
  Nausea and vomiting will be recorded if they occur after changing the infusion until the end of delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Jinjiang District Women & Children Health Hospital,, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
For our study "Effects of Different Concentrations of Ropivacaine on Prolonged Labor Analgesia," we have decided not to share Individual Participant Data (IPD). This decision is due to privacy concerns, data security requirements, ethical approval limitations, legal restrictions, and the study's design which did not accommodate data sharing. We believe this aligns with ethical standards and operational capabilities.

REFERENCES:
- [Result] Jian Z, Longqing R, Dayuan W, Fei J, Bo L, Gang Z, Siying Z, Yan G. Prolonged duration of epidural labour analgesia decreases the success rate of epidural anaesthesia for caesarean section. Ann Med. 2022 Dec;54(1):1112-1117. doi: 10.1080/07853890.2022.2067353. PMID 35443838
- [Result] Ni JX, Feng JL, Yao SJ, Ni LF, Song SB, Song CZ, Qian XW, Mei Z, Yu J. Determination of the Dose-Response Relationship of Epidural Dexmedetomidine Combined with Ropivacaine for Labor Analgesia. Drug Des Devel Ther. 2022 Mar 6;16:609-618. doi: 10.2147/DDDT.S346842. eCollection 2022. PMID 35281318
- [Result] Tan HS, Reed SE, Mehdiratta JE, Diomede OI, Landreth R, Gatta LA, Weikel D, Habib AS. Quality of Labor Analgesia with Dural Puncture Epidural versus Standard Epidural Technique in Obese Parturients: A Double-blind Randomized Controlled Study. Anesthesiology. 2022 May 1;136(5):678-687. doi: 10.1097/ALN.0000000000004137. PMID 35157756
- [Result] Hawkins JL. Epidural analgesia for labor and delivery. N Engl J Med. 2010 Apr 22;362(16):1503-10. doi: 10.1056/NEJMct0909254. No abstract available. PMID 20410515
- See also: Related Info — https://www.jjfck.com/